CLINICAL TRIAL: NCT00708539
Title: A Prospective Randomized Multicentre Study to Compare Crinone 8% Once Daily Versus Other Vaginal Progesterone.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordica Fertility Clinic (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Professor Svend Lindenberg, Nordica fertility clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25921; Eudra CT nr.2005-001248-22
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-07

CONDITIONS: IVF - Luteal Phase Support After Embryo Transfer
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Crinone vaginal gel 8% 90 mg once daily
  Interventions: Drug: progesterone
- 2 (Active Comparator): Progesterone mic 400 mg three times daily
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: progesterone — 90 mg, vaginal, once daily
  Other Names: crinone 8%
  Arms: 1
Drug: Progesterone — 200 mg, vaginal, three times daily used in Denmark, 400 mg, vaginal, three times daily used in Sweden
  Other Names: Progestan in Denmark; Progesterone mic in Sweden
  Arms: 2

SUMMARY:
To compare the effect of Crinone 8% administered once daily versus other vaginal progesterone in terms of ongoing pregnancy rate 5 weeks after embryo transfer as well as patient convenience.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Regular menstrual cyclus 25-35 days
* both ovaries present
* No more than 2 previous IVF attempts
* Have given written informed consent

Exclusion Criteria:

* More than 2 previous attempts
* Known drug abuse
* Known allergies to the study medication
* No embryo transfer performed in the study cycle
* Previous participating in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2686 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Equivalence in ongoing pregnancy per embryo transfer between the two groups | week 5 after embryo tranfer

SECONDARY OUTCOMES:
Convenience for the patient | the treatment period (from the day of embryo transfer and 19 days ahead)

CONTACTS AND LOCATIONS:
Overall Officials: Svend Lindenberg, Principal Investigator — Nordica Fertilityclinic; Svend Lindenberg, Principal Investigator — Nordica Fertility Clinic
Locations (17):
- Denmark (12):
  - Faurskov fertility clinic, Aalborg
  - Brædstrup Sygehus, Brædstrup
  - Dronninglund sygehus, Dronninglund
  - Dansk Fertilitetsklinik, Frederiksberg
  - Herlev Hospital, Herlev
  - Holbæk Sygehus, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Rigshospitalet, København Ø
  - Odense IVF, Odense
  - Odense OUH, Odense
  - Roskilde Sygehus, Roskilde
  - Skive sygehus, Skive
- Sweden (5):
  - Reproduktionscentrum, Sahlgrenska, Gothenburg
  - Karolinska, Huddinge
  - RMC, Malmo
  - Reproduktionscentrum, Stockholm
  - Norrlandsuniversitets sjukhus, Umeå